CLINICAL TRIAL: NCT00116311
Title: Effects of Allergen Inhalation on Adenosine Receptor Expression and Mast Cell Activation in Peripheral Blood and Sputum of Asthmatics and Healthy Subjects
Brief Title: Effects of Allergen Inhalation on Adenosine Receptor Expression in Sputum and Peripheral Blood
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Groningen Research Institute for Asthma and COPD (Other)
Other Study IDs: METc2004-253
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2007-03

CONDITIONS: Asthma; Healthy
Keywords: Adenosine receptors; asthma; sputum; peripheral blood; healthy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: allergen inhalation
Behavioral: withdrawal of medication
Procedure: sputum induction

SUMMARY:
The purpose of this study is to determine whether asthmatics have different adenosine receptor expression profiles than healthy controls. We hypothesize that asthmatics will have increased adenosine receptor expression versus control subjects.

We also want to study the effects of allergen inhalation on adenosine receptor expression in asthmatics. We believe that adenosine receptor expression will be upregulated after allergen inhalation.

Both hypotheses are being tested in sputum and peripheral blood.

ELIGIBILITY:
Asthmatic Subjects - Inclusion Criteria:

* Clinical diagnosis of asthma
* Steroid naive or subjects not using their inhaled steroids for the last 4 weeks, short-acting beta-agonist for rescue medication
* FEV1 > 70% of predicted
* Positive skin prick test for house dust mite, cat or grass pollen
* PC20 methacholine or histamine < 8 mg/ml

Asthmatic Subjects - Exclusion Criteria:

* Use of systemic steroids in the previous 6 weeks
* Asthma exacerbations in the previous 6 weeks
* Current or ex-smokers with ≥ 10 pack-years (≥ 2 pipe pack-years), ex smokers who stopped less than 1 year ago

Healthy Subjects - Inclusion Criteria:

* No airway complaints
* FEV1 > 90% of predicted
* Negative skin prick test
* PC20 methacholine or histamine > 8 mg/ml

Healthy Subjects - Exclusion Criteria:

* Use of steroids in the previous 6 weeks
* Current or ex-smokers with ≥ 10 pack-years (≥ 2 pipe pack-years), ex smokers who stopped less than 1 year ago

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-07; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Dirkje S Postma, prof. MD PhD, Principal Investigator — University Medical Center Groningen, Department of Pulmonology, hanzeplein 1, 9713 GZ Groningen, The Netherlands
Locations (1):
- University Medical Center Groningen, Department of Pulmonology, Groningen, Netherlands